CLINICAL TRIAL: NCT00690066
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of PROCHYMAL® (Ex Vivo Cultured Adult Human Mesenchymal Stem Cells) for the Treatment of Recently Diagnosed Type 1 Diabetes Mellitus
Brief Title: PROCHYMAL® (Human Adult Stem Cells) for the Treatment of Recently Diagnosed Type 1 Diabetes Mellitus (T1DM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mesoblast, Inc. (Industry)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 901
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Type 1 Diabetes Mellitus; Type 1 Diabetes; Diabetes Mellitus, Insulin-Dependent; Juvenile Diabetes
Keywords: T1DM; Type 1 Diabetes Mellitus; Type 1 Diabetes; Diabetes Mellitus, Insulin-Dependent; Juvenile Diabetes; Adult Human Stem Cells; Mesenchymal Stem Cells; MSCs; Insulin; Osiris; Prochymal
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — remestemcel-l

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prochymal (Experimental): PROCHYMAL®
  Interventions: Drug: PROCHYMAL®
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PROCHYMAL® — Intravenous infusion of ex vivo cultured adult human mesenchymal stem cells
  Other Names: ex vivo cultured adult human mesenchymal stem cells; Prochymal
  Arms: Prochymal
Drug: Placebo — Intravenous infusion of excipients of PROCHYMAL®
  Arms: Placebo

SUMMARY:
The purpose of this study is to establish the safety and efficacy of multiple administrations of PROCHYMAL® in participants recently diagnosed with type 1 diabetes mellitus.

DETAILED DESCRIPTION:
Diabetes mellitus refers to disorders in which the body has trouble controlling its blood glucose levels. There are two main types of diabetes: type 1 and type 2. Type 1 diabetes mellitus (T1DM), which is being studied in this trial, is an autoimmune disorder in which the body's own immune system attacks and destroys the cells that make insulin. These cells are called beta cells. As beta cells are destroyed, less insulin can be made. This causes blood sugar levels to increase above normal and can cause life-threatening hypo- and hyper-glycemic reactions. For this reason, people with type 1 diabetes must take insulin to help control their blood sugar levels. Over time, poorly controlled diabetes can lead to a variety of serious health conditions, including heart disease, stroke, blindness, amputations, kidney disease, and nerve damage. Insulin is the primary method of controlling diabetes by regulating blood glucose levels, but it may not reverse or prevent disease progression. The active ingredient in PROCHYMAL® is adult human mesenchymal stem cells (MSCs). MSCs have been shown to interact with the immune cells in the body, reducing inflammation and assisting in tissue repair. This study will help determine whether MSCs can protect normal pancreatic tissue from autoimmune attack and repair damaged pancreatic tissue, leading to an increase in insulin production and decrease in circulating blood glucose. The characteristics and biologic activity of PROCHYMAL®, along with a good safety profile in human trials to date, suggest that PROCHYMAL® may be a good candidate for addressing Type 1 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a diagnosis of type 1 diabetes mellitus based on the American Diabetes Association (ADA) criteria.
* Participant must be screened between 2 and 20 weeks from initial T1DM diagnosis
* Participants must be between the ages of 12 and 35 (inclusive).
* Participant must have at least one diabetes-related autoantibody present (either GAD or IA-2).
* Participant must have some beta cell function as determined by C-peptide testing (at least 0.2 pmol/mL (0.6 ng/mL) during MMTT.
* Participants must be willing to comply with "intensive diabetes management" as directed by the Investigator with the goal of maintaining blood glucose as close to normal as possible (i.e., glycosylated hemoglobin A1c (HbA1c) value of ≤ 7.0%).
* Participants must be willing to comply with the schedule of study visits and protocol requirements.

Exclusion Criteria:

* Participant has Body Mass Index (BMI) ≥ 30.
* Participant has evidence of retinopathy at baseline.
* Participant has abnormally high lipid levels.
* Participant has abnormal blood pressure.
* Participant has an abnormal serum creatinine.
* Participant has evidence of clinically significant proteinuria.
* Participant has diabetic ketoacidosis.
* Participant is being treated for a severe active infection of any type.
* A female participant who is breast-feeding, pregnant, or intends to become pregnant during the study.
* Participant with clinically relevant uncontrolled medical condition not associated with diabetes (e.g. hematologic, renal, hepatic, neurologic, cardiac, or respiratory).
* Participant has received an investigational drug (not approved by the FDA) for any indication 30 days prior to the screening visit.
* Participant is allergic to bovine or porcine products.
* Participant has evidence of active malignancy or prior history of active malignancy that has not been in remission for at least 5 years.
* Participant has any medical condition, which in the opinion of the Investigator, rendered his/her participation in this study unsuitable.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2008-06-11 (Actual); Primary Completion 2010-12-12 (Actual); Study Completion 2011-12-19 (Actual)

PRIMARY OUTCOMES:
C-peptide area under the concentration curve (AUC) response (MMTT) | 1 year

SECONDARY OUTCOMES:
Peak C-peptide response (MMTT) | 2 years
Basal C-peptide response | 2 years
Total daily insulin dose (units/kg) | 2 years
Glycosylated hemoglobin (HbA1c) levels | 2 years
Number of severe and documented hypoglycemic events | 2 years
Changes in levels of glutamic acid decarboxylase (GAD) or islet antigen 2 (IA-2) autoantibodies | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mahboob Rahman, MD, Study Director — Mesoblast, Inc.
Locations (20):
- United States (20):
  - University of Alabama, Division of Endocrinology & Metabolism, Birmingham, Alabama
  - Scripps Whittier Diabetes Institute, La Jolla, California
  - Stanford University, Stanford, California
  - University of Florida, Gainesville, Florida
  - Diabetes Research Institute, Miami, Florida
  - University of Kentucky, Lexington, Kentucky
  - University of Minnesota, Minneapolis, Minnesota
  - Desert Endocrinology CRC, Henderson, Nevada
  - Nevada Alliance Against Diabetes, Las Vegas, Nevada
  - University of North Carolina Diabetes Care Center, Chapel Hill, North Carolina
  - American Health Research, Inc., Charlotte, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - Providence Health Partners - Center for Clinical Research, Dayton, Ohio
  - Cumberland Valley Endocrinology, Carlisle, Pennsylvania
  - AM Diabetes & Endocrinology Center, Bartlett, Tennessee
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Optimum Clinical Research, Inc., Salt Lake City, Utah
  - The Strelitz Diabetes Center, Eastern VA Medical School, Norfolk, Virginia
  - University of Wisconsin Health- West Clinic, Madison, Wisconsin
  - Clinical and Transitional Science Institute, Milwaukee, Wisconsin